CLINICAL TRIAL: NCT02884128
Title: A Multi-Center, Open-Label Phase I Dose-Escalation Study of PEP02 in Combination With 5-fluorouracil (5-FU) and Leucovorin (LV) in Advanced Solid Tumors
Brief Title: A Study of PEP02 in Combination With 5-fluorouracil (5-FU) and Leucovorin (LV) in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP0203
Record Dates: First submitted 2016-08-12; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEP02 + 5-FU/LV (Experimental): The initial starting dose of PEP02 is 60 mg/m2, and was escalated by increments of 20 mg/m2 between dose levels. 5-FU and LV were given as 24-hour infusion via an implanted central venous catheter, with dose fixed at 2000 mg/m2 and 200 mg/m2, respectively. PEP02 was administered on Day 1; 5-FU/LV was started after the end of PEP02 infusion on Day 1 and also on Day 8.
  Interventions: Drug: PEP02; Drug: 5-FU; Drug: LV

INTERVENTIONS:
Drug: PEP02 — PEP02 was administered on Day 1. Treatment repeated every 3 weeks and it was regarded as one cycle of treatment.
  Other Names: liposomal irinotecan
Drug: 5-FU — 5-FU/LV were started after the end of PEP02 infusion on Day 1 and also on Day 8. Treatment repeated every 3 weeks and it was regarded as one cycle of treatment.
  Other Names: Fluorouracil
Drug: LV — 5-FU/LV were started after the end of PEP02 infusion on Day 1 and also on Day 8. Treatment repeated every 3 weeks and it was regarded as one cycle of treatment.
  Other Names: Leucovorin

SUMMARY:
This trial is a multi-center, open-label, phase I, dose escalation study of PEP02 (liposomal encapsulated irinotecan) in combination with 5-FU and LV in patients with advanced solid tumors.

DETAILED DESCRIPTION:
In this study, the initial starting dose of PEP02 is 60 mg/m2, and was escalated by increments of 20 mg/m2 between dose levels. 5-FU and LV was given as 24-hour infusion via an implanted central venous catheter, with dose fixed at 2000 mg/m2 and 200 mg/m2, respectively. PEP02 was administered on Day 1; 5-FU/LV was started after the end of PEP02 infusion on Day 1 and also on Day 8. Treatment repeated every 3 weeks and it was regarded as one cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor which was locally advanced or metastatic and had failed to standard chemotherapy or no standard treatment was available
* ECOG performance status 0 or 1
* With normal organ and marrow function

Exclusion Criteria:

* Have had major surgery, chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or have not recovered from toxicities due to previous treatment
* With known or suspicious primary or secondary brain tumors
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PEP02, 5-FU or leucovorin
* HBsAg+ or anti-HCV+ patients with splenomegaly (defined as spleen size > 11 cm in CT scan)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, and history of symptomatic congestive heart failure of Functional Class II or more (New York Heart Association) and ischemic heart diseases (i.e. myocardial infarction or angina pectoris), cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding females (a pregnancy test must be performed on all females who are of child-bearing potential before entering the study and the result must be negative)
* Had received irinotecan treatment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0 | 3 weeks

SECONDARY OUTCOMES:
objective tumor response according to Response Evaluation Criteria In Solid Tumours (RECIST) 1.0 | 6 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiang NJ, Chao TY, Hsieh RK, Wang CH, Wang YW, Yeh CG, Chen LT. A phase I dose-escalation study of PEP02 (irinotecan liposome injection) in combination with 5-fluorouracil and leucovorin in advanced solid tumors. BMC Cancer. 2016 Nov 21;16(1):907. doi: 10.1186/s12885-016-2933-6. PMID 27871319